CLINICAL TRIAL: NCT06982092
Title: Study of Effects of Neostigmine Versus Sugammadex in Ultrasonographic Evaluation of Recovery of Diaphragmatic Function After General Anesthesia
Brief Title: Using Diaphragm Ultrasonography, Sugammadex Recovers Diaphragmatic Function More Effectively Than Neostigmine.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU MS535/2024
Record Dates: First submitted 2025-04-04; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Perioperative Diaphragmatic Function
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Intervention Model Description: Interventional, parallel
Who Masked: Participant, Care Provider
Masking Description: double (Participant, Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sugammadex (Active Comparator): Group A: receive sugammadex (SUG group) as the reversal drug
  Interventions: Drug: sugammadex
- neostigmine (Active Comparator): receive neostigmine (NEO group) as reversal drug.
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: sugammadex — : patients will receive the reversal drug according to the group to which they had been randomised. in the Sugammadex Group will receive 2 mg/kg sugammadex.
  Other Names: bridion
  Arms: sugammadex
Drug: Neostigmine — Patients in the NEO Group will receive 50 mic/kg neostigmine and .01-.02 mg/kg atropine
  Arms: neostigmine

SUMMARY:
The aim of our study is to assess differences in the recovery of muscle function, using diaphragm ultrasonography, after reversal of a rocuronium-induced block, using neostigmine versus sugammadex

DETAILED DESCRIPTION:
Post-operative residual curarization (PORC) remains an essential clinical challenge. The possibility of assessing muscle function and excluding PORC using noninvasive tools in the perioperative period is very attractive. Therefore, we used diaphragm ultrasonography.

The diaphragm is a major respiratory muscle, accounting for 60-70% of the respiratory workload. Its dysfunction involves post-operative respiratory failure.

Diaphragm ultrasound imaging is a cheap and portable technique that allows assessment of diaphragm thickness, thickening, and excursion at a point in time or over time, in ambulatory patients and in mechanically ventilated patients.

Acetylcholinesterase inhibitors can reverse muscle block, but their short half-life may lead to residual curarization in the ward, especially when intermediate or long-acting NMBAs have been administered. Sugammadex is the first selective reversal drug for steroidal NMBAs; it has been shown to give full and rapid recovery of muscle strength, thus minimizing the occurrence of residual curarization.

This study was designed to assess differences in the recovery of the diaphragmatic function, using diaphragm ultrasonography, after reversal of a rocuronium-induced block, using neostigmine versus sugammadex.

It was conducted to 60 patients of both sexes, scheduled for FESS surgeries who underwent deep neuromuscular block with rocuronium. Cases were aged 18-65 years, ASA physical status ІІ or III.

The patients were randomized by computer software randomization and divided into two equal groups; SUG group (n =30 patients) that received 2 mg/kg sugammadex and NEU group (n =30 patients) that received 50 mic/kg and 0.01-0.02 mg/kg atropine.

The following parameters were assessed and recorded; diaphragmatic thickening fraction, diaphragmatic excursion, number of patient with baseline diaphragmatic functionat 30min, spirometry volume, post extubation heart rate, respiratory rate, saturation, bronchospasm, nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists' (ASA) physical status I or II or III
* Adult patients aging (18-65) years of both sexes. who undergoing deep neuromuscular block with rocuronium.
* Patients Scheduled for elective FISS surgery

Exclusion Criteria:

* Patient's refusal of procedure or participation in the study.
* ASA class IV.
* History of hepatic disease (Child Pugh B or C class).
* History of renal disease.
* Allergy or hypersensitivity to sugammadex or neostigmine.
* History of neuromuscular disease.
* Diaphragmatic palsy, pregnancy, nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
the difference between diaphragmatic thickening fraction at 30 minuets vs. The corresponding baseline values | By using diaphragmatic ultrasonography baseline diaphragmatic thickening fraction preoperative and at Zero time, 10 minutes, and 30 minutes in Post anesthesia care unit
  Prior to induction of anesthesia, baseline thickening fractioning evaluated using diaphragmatic ultrasonography, All patients were given general anesthesia, after pre-oxygenation induction of anesthesia was started using fentanyl and propofol. Intubation was done with proper size endotracheal tube after relaxation provided by rocuronium, At the end the operation patients received the reversal drug according to the group to which they had been randomised.
  Immediately prior to extubation, diaphragm ultrasonography was carried out to assess muscle recovery in each patient during spontaneous breathing. Two additional diaphragm ultrasound sessions were carried out 10 minutes and 30 minutes after discharge from the operating theatre, while the patients are in the post anesthesia care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Hamed Mahmoud, M.B.B.CH, Principal Investigator — Anesthesia resident Ain Shams University
Locations (1):
- faculty of medicine, ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: before 3/2025
Access Criteria: free